CLINICAL TRIAL: NCT01841918
Title: Phase II Safety and Immunogenicity of Live Attenuated Influenza H5 Candidate Vaccine Strain A/17/Turkey/Turkey/05/133 (H5N2) in Healthy Thai Volunteers
Brief Title: Safety and Immunogenicity of Live Attenuated Influenza H5N2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: The Government Pharmaceutical Organization (Other Government); World Health Organization (Other)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GPO AVIAN FLU Vaccine-V02-2
Record Dates: First submitted 2013-01-29; First posted 2013-04-29 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-07

CONDITIONS: Influenza Due to Influenza A Virus Subtype H5N2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A/17/turkey/Turkey/05/133 (H5N2) (Experimental): 100 participants will be admitted in the isolation ward for 5 days after each immunization mainly for safety assessment. Two doses of live attenuated influenza H5 vaccine candidate strain A/17/turkey/Turkey/05/133 (H5N2) will be given by intranasal route 28 days apart and will be followed for the total of 60 days.
  Interventions: Biological: Avian Flu Vaccine
- Placebo (Placebo Comparator): 50 participants will be admitted in the isolation ward for 5 days after each administered placebo mainly for safety assessment. Two doses placebo will be given by intranasal route 28 days apart and will be followed for the total of 60 days.
  Interventions: Biological: Avian Flu Vaccine

INTERVENTIONS:
Biological: Avian Flu Vaccine

SUMMARY:
The purpose of this study is to evaluate immune response and safety of live attenuated influenza H5 vaccine candidate strain A/17/turkey/Turkey/05/133 (H5N2) manufactured by GPO, Thailand in healthy Thais.

DETAILED DESCRIPTION:
It is a double blind randomized study using 7.5-8.5 log EID50 dose which is the same dose as being tested in phase I.

150 participants (100 vaccinees and 50 placebos) age 18-49 years old will be enrolled. All will be separated in 4 batches; Batch 1: 36 participants (24 vaccinees and 12 placebos) Batch 2: 38 participants (25 vaccinees and 13 placebos) Batch 3: 38 participants (25 vaccinees and 13 placebos) Batch 4: 38 participants (26 vaccinees and 12 placebos)

Each batch will be admitted in the isolation ward for 5 days after each immunization mainly for safety assessment. Two doses of live attenuated influenza H5 vaccine candidate strain A/17/turkey/Turkey/05/133 (H5N2) will be given by intranasal route 28 days apart. Total follow up is 60 day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 18-49 years old
* Having Thai ID card or equivalent
* Are seronegative to the specific H5 influenza virus determined by antibody titer less than 1:40 by HAI test to the corresponding antigen.
* Anti HIV - Negative
* All hematology, biochemistry and urine analysis are within normal range or of no clinical significance (not more than 1.5 times of normal value)
* Able to read and write and sign written informed consent.

Exclusion Criteria:

* Known history of egg allergy
* Having had recently influenza infection confirmed as H5
* History of bronchial asthma
* History of chronic lung diseases
* History of chronic rhinitis
* History of immunodeficiency state
* History of immunosuppression
* History of heavy smoking (more than 5 rolls per day)
* History of alcoholic (pure drink 200 ml per day)
* Acute infectious and noninfectious diseases (within 2 weeks)
* Exacerbation of chronic diseases or cancer or HIV positives
* Anamnestic leukocytosis, hepatitis B and C positives
* The volunteers who have been taking immunoglobulin products or have had a blood transfusion during past three months before the beginning of the experiment
* Participation in other research study or stop participant less than 1 month
* Pregnancy or plan to become pregnant for 60 days after enrollment or breast feeding
* Any concomitant medication with Aspirin
* Poultry workers

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Phase II safety and immunogenicity of live attenuated influenza H5 candidate vaccine strain A/17/turkey/Turkey/05/133 (H5N2) in healthy Thai volunteers | within 60 days after screening

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Tropical Medicine, Bangkok, Thailand

REFERENCES:
- [Derived] Pitisuttithum P, Boonnak K, Chamnanchanunt S, Puthavathana P, Luvira V, Lerdsamran H, Kaewkungwal J, Lawpoolsri S, Thanachartwet V, Silachamroon U, Masamae W, Schuetz A, Wirachwong P, Thirapakpoomanunt S, Rudenko L, Sparrow E, Friede M, Kieny MP. Safety and immunogenicity of a live attenuated influenza H5 candidate vaccine strain A/17/turkey/Turkey/05/133 H5N2 and its priming effects for potential pre-pandemic use: a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2017 Aug;17(8):833-842. doi: 10.1016/S1473-3099(17)30240-2. Epub 2017 May 19. PMID 28533093